CLINICAL TRIAL: NCT05117177
Title: A Multicenter, Open-Label, Phase I Clinical Study to Assess the Safety, Tolerability, Pharmacokinetics and Food-Effect of Inupadenant New Formulations in Participants with Advanced Solid Tumors
Brief Title: New Formulation Study of Inupadenant (EOS100850) in Patients with Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: iTeos Therapeutics (Industry)
Collaborators: iTeos Belgium SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A2A-004; 2020-005861-15 (EudraCT Number)
Record Dates: First submitted 2021-09-01; First posted 2021-11-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor, Adult
Keywords: Solid Tumor; Advanced Cancers; Phase I; Pharmacokinetics; Safety; Immunotherapy; Adenosine; Inupadenant

STUDY DESIGN:
Intervention Model Description: Arm 1: sequential dose escalation Arm 2: randomized crossover Arm 3: single treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Inupadenant sequential dose escalation (Part 1A) (Experimental): Part 1A will evaluate the safety as well as to determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of inupadenant in participants with advanced solid tumors.
  Interventions: Drug: Inupadenant
- Inupadenant randomized crossover (Part 1B) (Experimental): The effect of food on the exposure to inupadenant will be investigated in participants with advanced solid tumors.
  Interventions: Drug: Inupadenant
- Inupadenant single treatment assignment (Part 1C) (Experimental): Part 1C will investigate an additional formulation of inupadenant in participants with advanced solid tumors.
  Interventions: Drug: Inupadenant

INTERVENTIONS:
Drug: Inupadenant — Oral administration
  Other Names: EOS100850
  Arms: Inupadenant sequential dose escalation (Part 1A)
Drug: Inupadenant — Oral administration
  Other Names: EOS100850
  Arms: Inupadenant randomized crossover (Part 1B)
Drug: Inupadenant — Oral administration
  Other Names: EOS100850
  Arms: Inupadenant single treatment assignment (Part 1C)

SUMMARY:
A2A-004 is a three-part multicenter, open-label, Phase I clinical trial intended to evaluate the safety and tolerability, and the pharmacokinetics (PK) and food effect of new formulations of inupadenant (formerly known as EOS100850), in participants with advanced solid tumors.

ELIGIBILITY:
For more information regarding participation in the Trial, please refer to your physician

Inclusion Criteria:

* Women and men ≥18 years of age with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Subject with histologically or cytologically confirmed advanced solid tumor for whom no standard treatment is further available.
* At least 4 weeks since any previous treatment for cancer
* Subject must consent to pretreatment and on treatment tumor biopsies
* Adequate organ and marrow function

Exclusion Criteria:

* Patients with primary brain tumors or primary tumors with central nervous system metastases as only location of disease. Controlled brain metastases are permitted
* Participants with second/other active cancers requiring current treatment
* Uncontrolled/significant heart disease
* Known History of chronic hepatitis, Positive test for Hepatitis B virus surface antigen or - - Hepatitis C antibody (except participants with liver cancer) or Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome(HIV/AIDS)
* Active/uncontrolled autoimmune disease
* Active infection
* Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) in patients with advanced solid tumors receiving inupadenant | During the DLT evaluation period that is cycle 1 (each cycle is 4 weeks)
  Incidence of adverse events (AEs), serious adverse events (SAEs), DLTs, AEs leading to discontinuation, deaths, electrocardiogram (ECG) abnormalities, and clinically significant laboratory abnormalities
Incidence and severity of AEs in patients receiving inupadenant | Through study completion, an average of 4 months
  To assess safety and tolerability as measured by incidence and severity of AEs

SECONDARY OUTCOMES:
Plasma concentration of inupadenant vs. time profiles | Through study completion, an average of 4 months
  Determined by inspection of the concentration-time profile
Maximum observed serum concentration (Cmax) | Through study completion, an average of 4 months
  Determined by inspection of the concentration-time profile
Time of maximum observed concentration (Tmax) | Through study completion, an average of 4 months
  Determined by inspection of the concentration-time profile
Area under the concentration-time curve in 1 dosing interval [AUC(TAU)] | Through study completion, an average of 4 months
  Determined by inspection of the concentration-time profile
Plasma concentration half-life (T-HALF) | Through study completion, an average of 4 months
  Determined by inspection of the concentration-time profile
Overall response rate per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 | Through study completion, an average of 4 months
  Assessment of preliminary efficacy of inupadenant

CONTACTS AND LOCATIONS:
Overall Officials: Iteos Clinical Trials, Study Director — iTeos Belgium SA
Locations (5):
- Belgium (4):
  - GZA Ziekenhuizen, Wilrijk, Antwerpen
  - Cliniques Universitaires St-Luc, Brussels, Brussels Capital
  - University Hospital Ghent, Ghent, Ghent
  - Institut Jules Bordet, Anderlecht
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No